CLINICAL TRIAL: NCT03596008
Title: A Pilot Study Investigating the Effect of Acute Strawberry Intake on Endothelial Function Measured by Flow Mediated Dilation
Brief Title: Acute Strawberry Intake on Endothelial Function
Acronym: SFMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB2018-065
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: strawberry; monocytes; endothelial function

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, 2-arm, placebo-controlled, within subject cross-over trial, featuring a repeated postprandial sampling paradigm
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active1 (Experimental): freeze-dried strawberry powder (25 g) in active drink
  Interventions: Dietary Supplement: Active drink
- Placebo (Placebo Comparator): Placebo drink
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Active drink — The freeze-dried strawberry powder (25 g) in active drink
  Other Names: 25g strawberry drink
  Arms: Active1
Dietary Supplement: Placebo drink — Placebo drink
  Arms: Placebo

SUMMARY:
The primary objectives of the study are (1) to evaluate the effects of acute dietary strawberry intake on measures of vascular function in healthy adults following a meal challenge, (2) to evaluate the effects of acute dietary strawberry intake on metabolic status, and (3) to assess intervention-associated metabolite and inflammatory signatures and their relationship to vascular function.

DETAILED DESCRIPTION:
This study is a randomized, 2-arm, single-blinded, within subject cross-over trial focused on evaluating the effects of acute dietary strawberry intake on measures of vascular function, metabolic status, as well as metabolite and inflammatory signatures and their relationship to vascular function in healthy adults following a meal challenge.

A planned sample size of 15 will be enrolled into the study. This study will require one initial screening visit and 2 study visits. This study will take approximately 1 week per subject to complete.

The initial screening visit will provide subject with the informed consent document and determine subject eligibility through anthropometric measurements, vital signs, fasting blood glucose test (finger prick), and completion of a survey relate to general eating, health, and exercise habits.

If willing and eligible to participate, subjects will be invited to participate in the study for 2 study days. Subjects will be instructed to maintain their usual diet pattern and physical activity throughout study duration.

Subject will arrive at the center in a fasted state for at least 10 hours, well hydrated and rested. Each study visit will require blood draws and ultrasound measurement throughout the visit. After evaluation of subject's health status (via anthropometric, vital sign and blood glucose measurements and in-person interview), a Licensed Health Care Professional will place a catheter in subject's arm for the purpose of multiple blood sample collections and take the initial blood draw in the fasting state. A baseline FMD procedure will be completed immediately after baseline blood sample collection. Afterwards, subjects will be randomized to receive the strawberry powder treatment or placebo based on randomized treatment sequences for 2 study visits immediately after fasting blood draw. The sequences of receiving the supplement at each visit will be randomly assigned to one of 2 following sequences: A-B or B-A Each study visit will involve with blood samples collection at time points 0 (fasting), 1, 2, 4, 6, and 24 hour (h) for assessment of change in metabolites and inflammatory signatures. FMD procedure will be conducted after completing the baseline blood draw and later at 2h, 4h, 6h, and 24h. A standard breakfast will be provided immediately after the 0h blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 20 to 35 kg/m2
* Aged 18-45 years old
* Willing to maintain stable body weight and follow his/her habitual diet and physical activity patterns throughout the trail
* Judged by the Investigator to be in general good health on the basis of medical history and screening laboratory tests
* Able to provide informed consent and comply with study procedures

Exclusion Criteria:

* Current smoker and/or marijuana user, past smokers may be allowed in the study if stopped >2 years
* Have a history or presence of atherosclerotic cardiovascular disease, inflammatory disease, diabetes mellitus, or other systemic diseases, psychological or psychiatric disorders that may interfere with study outcomes
* Men and women with known or suspected intolerance, allergies or hypersensitivity to study foods or treatments
* Taking any medications and/or supplements that would interfere with outcomes of the study (i.e., lipid-lowering medications, anti-inflammatory drugs, etc),
* Unstable use of any medication/supplement
* Have a history of cancer, except for non-melanoma skin cancer within past 5 years
* Addicted to drugs and/or alcohol (>4 drinks/day)
* Have been exposed to any non-registered drug product within last 30 days.
* Working overnight (e.g. 3rd shift of overnight workers)
* Excessive exercisers or trained athletes
* Have allergies/intolerances to strawberries
* Extreme dietary habits (ie. vegetarian/vegan)
* Excessive coffee/tea drinker (>4 cups/day)
* Actively losing weight/ trying to lose weight (unstable body weight fluctuations of > 5 kg in 3 months)
* Donated blood within last 3 months
* Female who is pregnant, planning to be pregnant, breastfeeding
* Current regular consumption of berries which exceeds > 2 servings per day
* Any condition the Investigator believes would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.
* Fasting glucose concentration >125 mg/dL

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Changes in postprandial endothelial function using Flow Mediated Dilation (FMD) between 2 treatments | Baseline to 6 hours
  postprandial endothelial function using Flow Mediated Dilation (FMD)

SECONDARY OUTCOMES:
Change in plasma blood glucose concentration response between 2 treatments | Baseline to 24 hours
  blood glucose concentration response
Change in plasma blood insulin concentration response between 2 treatments | Baseline to 24 hours
  blood insulin concentration response

OTHER OUTCOMES:
Changes in plasma polyphenol metabolites between 2 treatments | Baseline to 24 hours
  plasma polyphenol metabolites
Changes in plasma inflammation (monocytes isolation) responses between 2 treatments | Baseline to 24 hours
  Monocytes inflammation responses

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No